CLINICAL TRIAL: NCT04857307
Title: A Multicenter, Open-Label Study to Evaluate the Pharmacokinetics, Tolerability, and Safety of a Single Dose of Staccato Alprazolam in Adolescent Study Participants With Epilepsy
Brief Title: A Study to Assess the Pharmacokinetics (PK) and Safety of Staccato Alprazolam in Adolescent Study Participants With Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0100
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Staccato alprazolam; Phase 1; Adolescents; STAP-001; Alprazolam
MeSH Terms: conditions — Epilepsy | interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Staccato alprazolam (Experimental): The study participants will receive a single dose of Staccato alprazolam.
  Interventions: Drug: Alprazolam

INTERVENTIONS:
Drug: Alprazolam — * Pharmaceutical form: Inhalation powder.
  * Study participants will receive Staccato alprazolam at prespecified time-points.
  Other Names: UCB7538

SUMMARY:
The purpose of the study is to assess the pharmacokinetics (PK), tolerability, and safety of Staccato alprazolam in adolescent study participants with epilepsy following single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 12 to 17 years of age inclusive, at the time of signing the Informed Consent form (ICF) and the Assent form
* Participant has an established diagnosis of focal, generalized, or focal and generalized epilepsy
* Participant is in good general health as determined by medical evaluation including medical history and physical examination
* Participants with a body weight ≥29 kg and body mass index (BMI) within the range 14 to 32 kg/m^2 (inclusive)
* A male participant must agree to use contraception
* A female participant is eligible to participate if she is not pregnant
* Participant is capable of and provides assent, and the study participant's parent/legal representative provides signed informed consent for minor study participants, which includes compliance with the requirements and restrictions listed in the ICF, Assent form, and in this protocol
* Participant has a lifetime history of never smoking >5 cigarettes/day, and a current history (for at least 6 months prior to Screening Visit) of not smoking at all (including e-cigarette and vaping products)
* Participant has forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) >80% predicted at Screening. In case of an out-of-range result, 1 repeat test will be allowed. If the readings are out-of-range again, the study participant will be excluded
* Participant is willing and able to be confined to a clinical research facility for up to 36 hours (including 1 overnight stay) and comply with the study schedule and study requirements.

Note: If there are no clinical contraindications, as per Investigator's judgment, study participants may leave the clinical research facility after the 6-hour postdose assessments and return to the clinic on Day 2 for the 24-hour and 36-hour postdose assessments

* Participant is currently taking at least 1 background antiepileptic drug (AED)
* Participant is able to actuate the training device during Screening, according to Instructions for Use

Exclusion Criteria:

* Participant has history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, neurological, hematological, cerebrovascular, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of Investigational Medicinal Product (IMP); constituting a risk when taking the study intervention; or interfering with the interpretation of data in the opinion of the Investigator
* Participant has a known hypersensitivity to any components of the IMP or comparative drugs (and/or an investigational device) as stated in the protocol
* Participant has severe chronic cardio-respiratory disease
* Participant has history of acute narrow angle glaucoma, hydrocephalus, or Myasthenia Gravis
* Participant has history or has current airway disease such asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* Participant has any acute respiratory signs/symptoms (ie, wheezing) and active acute respiratory infection (or within 1 week of dosing) with exception of symptoms of mild rhinitis
* Participant has a known hypersensitivity to albuterol or similar short-acting beta2-agonist (SABA) that may be used as rescue medication administered in response to potential bronchospasm
* Participant is taking strong liver inducing agents (eg, phenytoin, phenobarbital, carbamazepine, and primidone) or strong Cytochrome P450 3A4 (CYP3A4) inhibitors
* Participant has a SpO2 measured by pulse oximetry <95% for >30 seconds during the Screening Visit

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) following single inhaled dose of Staccato alprazolam | Plasma samples will be taken on Day 1 of the Treatment Period, predose and then following administration of Investigational Medicinal Product (IMP) at 2 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, and 36 hours postdose.
  Cmax = Maximum plasma concentration.
Area under the plasma concentration-time curve from zero to the last quantifiable concentration (AUC(0-t)) following single inhaled dose of Staccato alprazolam | Plasma samples will be taken on Day 1 of the Treatment Period, predose and then following administration of Investigational Medicinal Product (IMP) at 2 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, and 36 hours postdose.
  AUC(0-t) = Area under the plasma concentration-time curve from zero to the last quantifiable concentration.
Area under the plasma concentration-time curve from time 0 to infinity (AUC) following single inhaled dose of Staccato alprazolam | Plasma samples will be taken on Day 1 of the Treatment Period, predose and then following administration of Investigational Medicinal Product (IMP) at 2 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, and 36 hours postdose.
  AUC = Area under the plasma concentration-time curve from time 0 to infinity.
Apparent total body clearance (CL/F) following single inhaled dose of Staccato alprazolam | Plasma samples will be taken on Day 1 of the Treatment Period, predose and then following administration of Investigational Medicinal Product (IMP) at 2 minutes, 10 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 24 hours, and 36 hours postdose.
  CL/F = Apparent total body clearance.
Percentage of participants with treatment-emergent adverse event (TEAEs) | From baseline (Day 1) till end of Safety Follow-up (up to Day 9)
  An Adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant temporally associated with the use of IMP, whether or not considered related to the IMP.
Percentage of participants with serious treatment-emergent adverse event (serious TEAEs) | From baseline (Day 1) till end of Safety Follow-up (up to Day 9)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  a. Results in death c. Requires inpatient hospitalization or prolongation of existing hospitalization d. Results in persistent disability/incapacity e. Is a congenital anomaly/birth defect f. Important medical events.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (8):
- United States (8):
  - Up0100 102, Little Rock, Arkansas
  - Up0100 110, Orlando, Florida
  - Up0100 103, Honolulu, Hawaii
  - Up0100 101, Bethesda, Maryland
  - Up0100 108, Rochester, New York
  - Up0100 106, Cincinnati, Ohio
  - Up0100 105, Memphis, Tennessee
  - Up0100 107, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.